CLINICAL TRIAL: NCT06887738
Title: A Proof-of-Concept Phase II, Open-Label Study of NM8074 in Patients with Dermatomyositis (DM)
Brief Title: Study of NM8074 in Patients with Dermatomyositis (DM)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NovelMed Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NM8074-DM-701
Record Dates: First submitted 2025-03-07; First posted 2025-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Intervention Model Description: The proposed trial in DM subjects is designed as an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 1 (Experimental): All subjects will be administered 20 mg/kg of NM8074 intravenously every week, for a total of 12 doses from Day 1 to Day 78 of the treatment Period.
  Interventions: Drug: NM8074

INTERVENTIONS:
Drug: NM8074 — NM8074 will be administered as an intravenous infusion at a dose of 20mg/kg

SUMMARY:
This is a Phase II, open-label, multicenter study to evaluate the safety and efficacy of NM8074 administered via intravenous infusion in patients with Dermatomyositis (DM).

DETAILED DESCRIPTION:
The Proposed Study, NM8074-DM-701 will enroll a planned number of eight (8) DM subjects, with the potential to enroll more patients. The total duration of the study for all subjects will include a 30-day screening period, dosing for a 12-week Treatment Period, followed by an observation period of 6-weeks. All subjects will be administered 20 mg/kg of NM8074 intravenously every week for a total of 12 doses from Day 1 to Day 78 of the Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years of age at the time of consent.
* A body mass index (BMI) within the range of 15 - 38 kg/m2. BMI = Body weight (kg) / [Height (m)]2.
* Subjects diagnosed with a probable or definite DM according to 2017 European League Against Rheumatism/American College of Rheumatology (2017 EULAR/ACR).
* Subjects must have proof of vaccination against Neisseria meningitidis (MenACWY and MenB), Streptococcus pneumoniae (PCV13 or PCV15 and PPSV23), and Haemophilus influenzae type b (Hib) taken at least 2 weeks prior to NM8074 administration as per national and local guidelines. If the window of vaccination is short, then patients will be prophylactically treated with appropriate antibiotics.
* Female partners of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must have a negative pregnancy test at screening and must agree to use highly effective methods of contraception during dosing and for at least 8 weeks after stopping the investigational drug.
* Male patients and partners of child-bearing potential must agree to use contraceptives, and male patients must agree to refrain from donating sperm for the duration of the study and for at least 8 weeks after stopping the investigational drug.

Exclusion Criteria:

* Subjects with drug-induced myositis
* Subjects who have interstitial lung disease requiring the use of supplemental oxygen.
* Use of other investigational drugs at the time of enrollment, or within 5 half- lives of enrollment or within 3 months to study day 1, whichever is longer.
* History of currently active or suspicion of active bacterial, viral, or fungal infection within 2 weeks prior to first dose, or history of unexplained, recurrent bacterial infections.
* Subjects currently or previously diagnosed with cancer or who finished their cancer treatment within 2 years of the start of the clinical trial.
* Subjects with the history of bone marrow, hematopoietic stem cells, or solid organ transplantation.
* Has a currently active or known history of meningococcal disease or N. meningitidis infection.
* Evidence of active malignant disease or malignancies diagnosed within the previous 5 year
* Clinically significant medical or psychological conditions or risk factors that, as per the Investigator's judgment, could hinder the patient's participation in the study, introduce additional risks for the patient, or complicate the evaluation of the patient or study outcomes.
* Pregnant, planning to become pregnant, or nursing female subjects.
* Females with a positive pregnancy test result at Screening or on Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline or Percent Change from Baseline in the number of patients whose Total Improvement Score (TIS) has increased by ≥ 20 | Up to Study Day 78
  TIS is a composite measure used in clinical trials that integrates the 6 Core Set Measures (CSM). TIS scores range from 0-100, with 0-19, 20-39, 40-59, and 60-100 indicating no improvement, minimal, moderate, and major improvement respectively.

SECONDARY OUTCOMES:
Change from baseline or Percent Change from Baseline in Cutaneous Dermatomyositis Area and Severity Index (CDASI) score | Up to Study Day 78
  In DM, CDASI is a visual tool for a physician to assess the activity and damage of skin involvement in DM patients. The total activity score ranges from 0 to 100, and the damage score ranges from 0 to 32, wherein both criteria the higher score indicates more severe activity or damage of the disease in the patient.
Change from Baseline or Percent Change from Baseline in Manual Muscle Testing (MMT-8) parameter | Up to Study Day 78
  In Manual Muscle testing (MMT-8) eight specific muscle groups strengths are evaluated, each muscle group is scored on a scale from 0 (no movement) to 10 (normal strength), resulting in a maximum total score of 150 with a higher score indicating better muscle strength. Where a score < 136 would indicate muscle weakness significant enough to classify the patient as at risk of DM. MMT-8 can contribute between 0 to 32.5 points to the TIS: If there is a significant improvement in the patient's condition of more than 30% from baseline, the maximum score of 32.5 points is awarded. If the condition worsens or shows only a slight improvement (up to 2% from baseline), then 0 points are given.
Change from Baseline or Percent Change from Baseline in Physician's Global Activity (PhGA) assessment | Up to Study Day 78
  The PhGA is scored on a scale from 0 (no evidence of disease activity) to 10 (extremely severe disease), with higher scores indicating greater disease severity.
Change from Baseline or Percent Change from Baseline in Patient's Global Activity (PtGA) assessment | Up to Study Day 78
  The PhGA is scored on a scale from 0 (no evidence of disease activity) to 10 (extremely severe disease), with higher scores indicating greater disease severity.
Change from Baseline or Percent Change from Baseline Health Assessment Questionnaire (HAQ) score | Up to Study Day 78
  HAQ can contribute between 0 to 10 points to the TIS:
  - If there is a significant improvement in the patient's condition of more than 40% from baseline, the maximum score of 10 points is awarded. If the condition worsens or shows only a slight improvement (up to 5% from baseline), then 0 points are given.
Change from Baseline or Percent Change from Baseline in Extra muscular Activity (MDAAT) score | Up to Study Day 78
  Extra-muscular Activity can contribute between 0 to 20 points to the TIS:
  - If there is a significant improvement in the patient's condition of more than 40% from baseline, the maximum score of 20 points is awarded. If the condition worsens or shows only a slight improvement (up to 5% from baseline), then 0 points are given.

OTHER OUTCOMES:
Assessment for the presence of myositis-specific autoantibodies (MSA) | Up to Study Day 127
Change from Baseline or Percent Change from Baseline in Classical Pathway (CP) modulation | Up to Study Day 127
  NM8074-mediated CP inhibition is measure via a complement CP ELISA-based assay measuring MAC formation.
Change from Baseline or Percent Change from Baseline in plasma concentration of NM8074 | Up to Study Day 127
Maximum plasma concentration (Cmax) | Up to Study Day 127
Time corresponding to Cmax (tmax) | Up to Study Day 127
Area under the drug concentration-time curves (AUC0-t) | Up to Study Day 127

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lundberg IE, Tjarnlund A, Bottai M, Werth VP, Pilkington C, Visser M, Alfredsson L, Amato AA, Barohn RJ, Liang MH, Singh JA, Aggarwal R, Arnardottir S, Chinoy H, Cooper RG, Danko K, Dimachkie MM, Feldman BM, Torre IG, Gordon P, Hayashi T, Katz JD, Kohsaka H, Lachenbruch PA, Lang BA, Li Y, Oddis CV, Olesinska M, Reed AM, Rutkowska-Sak L, Sanner H, Selva-O'Callaghan A, Song YW, Vencovsky J, Ytterberg SR, Miller FW, Rider LG; International Myositis Classification Criteria Project consortium, The Euromyositis register and The Juvenile Dermatomyositis Cohort Biomarker Study and Repository (JDRG) (UK and Ireland). 2017 European League Against Rheumatism/American College of Rheumatology classification criteria for adult and juvenile idiopathic inflammatory myopathies and their major subgroups. Ann Rheum Dis. 2017 Dec;76(12):1955-1964. doi: 10.1136/annrheumdis-2017-211468. Epub 2017 Oct 27. PMID 29079590
- See also: Related Info — https://doi.org/10.1136/annrheumdis-2017-211468